CLINICAL TRIAL: NCT03325400
Title: In Vivo Comparison of Genotoxic and Cytotoxic Effects of Different Brands of Toothpaste - Without and With Fluoride
Brief Title: Cytogenetic Damage in Buccal Cells Caused by Toothpaste
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Split, School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Screening
Other Study IDs: USplitSM
Record Dates: First submitted 2017-10-20; First posted 2017-10-30 (Actual); Last update posted 2017-10-30 (Actual); Status verified 2017-10

CONDITIONS: Toxicity
Keywords: Fluoride toothpaste; Cytogenetic damage; Exfoliated buccal cells; Micronucleus assay
MeSH Terms: interventions — Fluorides; halofantrine

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Non-fluoride toothpaste (Other): Participants have used toothpaste for four months. The first two months they used non-fluoride toothpaste, after which, for the next two months, they used toothpaste containing fluoride of the same manufacturer and similar composition. The tested kinds of toothpaste were applied twice a day, in the morning and evening, for three minutes in the amount of 1 g (≈2 cm). Contemporary, participants did not use other agents for oral hygiene such as mouthwash or topical fluoridation.
  Interventions: Other: Toothpaste non-fluoride and fluoride
- Fluoride toothpaste (Active Comparator): Participants have used toothpaste for four months. The first two months they used non-fluoride toothpaste, after which, for the next two months, they used toothpaste containing fluoride of the same manufacturer and similar composition. The tested kinds of toothpaste were applied twice a day, in the morning and evening, for three minutes in the amount of 1 g (≈2 cm). Contemporary, participants did not use other agents for oral hygiene such as mouthwash or topical fluoridation.
  Interventions: Other: Toothpaste non-fluoride and fluoride

INTERVENTIONS:
Other: Toothpaste non-fluoride and fluoride — Participants have used toothpaste for four months. The first two months they used non-fluoride toothpaste, after which, for the next two months, they used toothpaste containing fluoride of the same manufacturer and similar composition. The tested kinds of toothpaste were applied twice a day, in the morning and evening, for three minutes in the amount of 1 g (≈2 cm).
  Participants have used toothpaste for four months. The first two months they used non-fluoride toothpaste, after which, for the next two months, they used toothpaste containing fluoride of the same manufacturer and similar composition. The tested kinds of toothpaste were applied twice a day, in the morning and evening, for three minutes in the amount of 1 g (≈2 cm). Contemporary, participants did not use other agents for oral hygiene such as mouthwash or topical fluoridation.
  Other Names: Sensodyne Classic (GlaxoSmithKline, UK), Sensodyne Fluor (GlaxoSmithKline, UK), Plidenta 15 Seconds (Neva Ltd., Croatia), Plidenta Sensitive (Neva Ltd., Croatia)

SUMMARY:
Objectives. Toothpaste contains many potentially harmful ingredients, including some that can lead to serious long-term health problems. Everyday use of oral health care products has increased, highlighting the need for healthcare clinicians and consumers to be informed of the potential benefits and risks associated with these products. The aim of this study is to evaluate possible DNA damages to oral epithelial cells in participants exposed to toothpaste containing fluoride as opposed to the effects of non-fluoride toothpaste.

Materials and Methods. Forty volunteers were selected among students of dental medicine and assigned into two experimental groups. Each group used regular non-fluoride toothpaste for initial two months, followed by the use of fluoride toothpaste of the same brand for the next two months. The buccal epithelial cells were sampled at baseline and 30, 60, 90 and 120 days after the beginning of the research. Chromosomal damages were analyzed by micronucleus assay.

DETAILED DESCRIPTION:
The study included 40 participants, students of Dental Medicine at the School of Medicine, of the University of Split. There were a total of 12 males and 28 females, aged between 20 and 26 (mean age 23.18 ± 1.48). Subjects were divided into two equal groups, depending on the combination of the toothpaste used.

In the first group, Sensodyne Classic (GlaxoSmithKline, UK) and Sensodyne Fluor (GlaxoSmithKline, UK) were the brands of toothpaste used, while in the second Plidenta 15 Seconds (Neva Ltd., Croatia) and Plidenta Sensitive (Neva Ltd., Croatia) (Table 1). Participants have used toothpaste for four months. The first two months they used non-fluoride toothpaste, after which, for the next two months, they used toothpaste containing fluoride of the same manufacturer and similar composition. The tested kinds of toothpaste were applied twice a day, in the morning and evening, for three minutes in the amount of 1 g (≈2 cm). Contemporary, participants did not use other agents for oral hygiene such as mouthwash or topical fluoridation. A detailed medical and dental anamnesis were taken from each participant. In a structured questionnaire, tailored to this study all participants provided answers to questions related to demographic factors (age, gender), personal factors (general health, a medication used, radiation exposure), lifestyle (smoking, alcohol consumption) eating habits and oral hygiene habits. Individuals who smoked three or more cigarettes a day for at least a year were considered as smokers. Those individuals who consumed two or more alcohol units for three or more times a week were not included in the study as well as patients with oral lesions, history of malignancy, and those with removable and fixed prosthodontics, orthodontic appliances. The criterion for selecting participants was to be completely healthy with no systemic disorders and diseases.

Sample collection Samples of buccal epithelial cells were collected from each participant using the swab technique immediately prior to the use of tested toothpaste and 30, 60, 90 and 120 days after the beginning of the research (T0 - control prior to the use of tested toothpaste, T1- 30 days after the beginning of the use of non-fluoride toothpaste, T2 - 60 days after the beginning of the use of non-fluoride toothpaste, T3 - 90 days after the beginning of the study, using fluoride toothpaste for 30 days, T4 - 120 days after the beginning of the study, using fluoride toothpaste for 60 days).

One hour prior the sampling, the participants were asked to abstain from smoking and consuming any food and drinks. After rinsing of the oral cavity for three times with tepid water in order to remove exfoliated cells, a swab was taken by gently brushing the buccal mucosa bilaterally with a cytobrush (Cytobrush Plus, GmbH, Dietramszell-Linden, Germany) and then the samples were applied to coded laboratory glass slides pre-warmed at 37 °C.

Micronucleus assay in buccal epithelial cells The cells applied on microscopic slides were allowed to air-dry and then were fixed in methanol (80% v/v) at 4°C for 20 minutes. Staining was carried out with 5% Giemsa solution for 10 minutes. Afterwards, the slides were rinsed with aqua distillate and air-dried.

The analysis was done under a light microscope Olympus CX40 (Olympus, Tokyo, Japan) with a 400× magnification, and each micronucleus and other nuclear anomalies were additionally verified under 1000× magnification. Two replicate slides were prepared for each subject, and 1000 epithelium cells per preparation were scored for each sampling time.

Statistical analysis Statistical analysis was done by using SPSS software package (IBM Corp., Armonk, NY, USA). By descriptive statistical analysis, the basic statistical parameters (mean, standard error, and standard deviation, and relative standard deviation, median and minimum and maximum values) were determined. The differences in the number of micronuclei and other nuclear anomalies between different sampling times for each group and between the groups of examinees were tested by ANOVA and Tukey's HSD post hoc test using a general linear model procedure. General regression model (GRM) from linear/nonlinear modelling method was used for the assessment of the influence of the predictor variables (age, gender, and profession, use of medication, X-ray exposure, dietary habits, and lifestyle) onto dependent variables (micronucleus, binucleated cells, broken eggs, nuclear buds, pyknosis, condensed chromatin, karyolysis and karyorrhexis). The results of GRM are expressed in the form of Pareto charts of t values. A significance level was set at 0.05.

ELIGIBILITY:
Inclusion Criteria:

* completely healthy (no systemic disorders and diseases)

Exclusion Criteria:

* consuming two or more alcohol units for three or more times a week
* patients with oral lesions
* history of malignancy
* patients with removable and fixed prosthodontics, orthodontic appliances.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2016-01-01 (Actual); Primary Completion 2016-06-15 (Actual); Study Completion 2016-07-20 (Actual)

PRIMARY OUTCOMES:
Cytogenetic damage | four months
  The aim of this study was to assess the number of buccal epithelial cells with cytogenetic defects in participants using commercial toothpaste with and without fluoride of the same manufactures and similar composition. Using the micronucleus assay, the effect of toothpaste on the buccal cells was monitored, depending on the time of the exposure.

IPD SHARING:
Plan to Share IPD: No
The data from individual respondents will not be available to other researchers

REFERENCES:
- [Background] Tadin A, Gavic L, Zeravica A, Ugrin K, Galic N, Zeljezic D. Assessment of cytotoxic and genotoxic effects of conventional and whitening kinds of toothpaste on oral mucosa cells. Acta Odontol Scand. 2018 Jan;76(1):64-70. doi: 10.1080/00016357.2017.1384567. Epub 2017 Sep 29. PMID 28959909